CLINICAL TRIAL: NCT07138469
Title: Overview of Elective Oocyte Preservation Three Years After Its Authorization in France: a Nationwide Multicenter Study
Brief Title: FRench Elective Oocyte prEservation: a Multicenter Study thrEe Years Later
Acronym: FREEZE-FR
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: BRUGNON_2023_CF094
Record Dates: First submitted 2025-06-25; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Elective Fertility Preservation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- women engaged in an elective fertility preservation process: women engaged in an elective fertility preservation process and who agree to participate in the study by completing the questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire was offered on a voluntary basis and completed online by the participants. At the end of the inclusion period, the responses were analyzed. Participant indicated in the questionnaire whether or not they had already undergone oocyte cryopreservation. The responses were analyzed to assess demographic characteristics, the level of knowledge regarding the bioethics law on non-medical fertility preservation, and future perspectives in the event of use (desired parental model, likelihood of use) or non-use.
  Other Names: Questionnaire developed by the AMP-CECOS unit of the Clermont-Ferrand University Hospital and approved by the ART unit team.

SUMMARY:
Previously reserved for pathological cases, oocyte cryopreservation for non-medical reason also named elective fertility preservation (EFP) is now authorized in France for women aged 29 to 37 following the revision of the bioethics law on August 2nd 2021. Currently, French data related to this new practice are lacking. The aim of this study is to conduct a preliminary assessment 3 years after approval of elective oocyte cryopreservation in France, evaluating the knowledge and perspectives of women undergoing elective fertility preservation in order to gain a better understanding of this new population and define the socio-economic and demographic profiles to improve care quality.

DETAILED DESCRIPTION:
This is a multicenter descriptive study conducted by the AMP-CECOS unit of the Clermont-Ferrand University Hospital between November 2023 and June 2024, with the participation of CECOS centers across mainland France. This national survey is carried out using an anonymous online questionnaire (Google Forms) developed at ART unit of Clermont Ferrand University Hospital and approved by the entire clinico-biological team. The study was submitted for ethical approval and compliance with the General Data Protection Regulation (GDPR) and received a favorable opinion from the Ethics Committee of the Clinical Research and Innovation Department (DRCI) of the Clermont-Ferrand University Hospital on July 24, 2023. The project was also presented to the scientific committee of the CECOS federation and published on two national reference platforms for fertility. Then, an envelope containing 50 flyers along with an explanatory note was sent by post to the 31 CECOS centers in mainland France.

Included in this study were women in a fertility preservation process for non-medical reasons, who have been seen in consultation as part of a request for non-medical fertility preservation, as well as women who have already undergone non-medical fertility preservation in France since its authorization on August 2, 2021. The inclusion criteria were those applicable to non-medical fertility preservation, being between 29 and 37 years of age at the time of care and not meeting the criteria for fertility preservation for medical reasons. An anonymous questionnaire using the Google Forms tool was elaborated by myself and approved by the clinico-biological team of the AMP-CECOS unit at the Clermont-Ferrand University Hospital. The survey takes only a few minutes to complete. It consisted of 18 questions, including open-ended (O), single-choice (SCQ), and multiple-choice (MCQ) questions. For most questions, a response was not mandatory to proceed with the questionnaire, in case participants prefer not to answer. To access the online survey, a flyer was prepared in advance and given to participants during their consultation. It includes the address https://bit.ly/enquete.fertilite and a QR code linking to the survey. A digital version was also sent by email to women who have already undergone oocyte cryopreservation. Three main themes emerged from the questionnaire. The first concerned the socio-economic and demographic data of the study population: department of residence, age, family status, parenthood, and level of education (SCQ). The second concerned the knowledge of the bioethics law governing the EFP (SCQ) and gamete donation (SCQ) and the third concerned the perspectives of participants for the use of cryopreserved oocytes (MCQ) and in case of non-use (MCQ).

ELIGIBILITY:
Inclusion Criteria:

* Being in SFP process
* Undergone SFP
* 29 to 37 years of age at the time of SFP or process

Exclusion Criteria:

* Women who had criteria for medical fertility preservation

Ages: 29 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women engaged in an elective fertility preservation process and who agree to participate in the study by completing the questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire to better define the demographic characteristics, knowledge, and perspectives of women who have undergone or wish to undergo oocyte cryopreservation for non-medical reasons. | 7 months (01/11/2023 to 30/06/2024)
  Department of residence, age group, stage of process, family status, marital status, education level, motivation, sources of information, knowledge of limit age for oocyte use, probability of use, perspectives of using cryopreserved oocytes: intended family model, perspectives in case of non-use of cryopreserved oocytes, knowledge of the bioethics law on the right of access to origins governing gamete donation

SECONDARY OUTCOMES:
Analysis of questionnaire responses based on whether or not fertility preservation has been performed, to assess the impact of the care stage on knowledge of the bioethics law. | 7 months (01/11/2023 to 30/06/2024)
  The investigators will examined whether there were differences in knowledge responses depending on whether fertility preservation had been carried out or not, and whether the women had already attended a consultation or not.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Dufaure, MD, Principal Investigator — University Hospital, Clermont-Ferrand; Florence Brugnon, MD,PhD,HDR, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: Undecided